CLINICAL TRIAL: NCT03353428
Title: Interventional Treatment of Lung Cancer (LC) With LC Specific Immune Lymphocytes (LC-CTLs)
Brief Title: Intervention of Engineered Immune Effector T Cells Against Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: combine with NCT03356808
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17022
Record Dates: First submitted 2017-11-20; First posted 2017-11-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer; NSCLC
Keywords: Lung cancer; Cytotoxic lymphocyte; LC-CTL; NSCLC
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LC-CTLs (Experimental): Autologous lung cancer specific cytotoxic lymphocytes
  Interventions: Biological: LC-CTLs

INTERVENTIONS:
Biological: LC-CTLs — 2 to 4 infusions, once a week, for 1x10^5~4x10^6 CTLs/kg via IV, chest or tumor injection each time

SUMMARY:
The primary objective of this study is to evaluate the safety of lung cancer specific cytotoxic lymphocytes (LC-CTLs). The secondary objectives are to evaluate the rate of successful LC-CTLs generation in vitro and determine the anti-lung cancer efficacy.

DETAILED DESCRIPTION:
Lung cancer is a malignant lung tumor characterized by uncontrolled cell growth in tissues of the lung. The two main types are small-cell lung carcinoma (SCLC) and non-small-cell lung carcinoma (NSCLC). Worldwide in 2012, lung cancer occurred in 1.8 million people and resulted in 1.6 million deaths. Common treatments include surgery, chemotherapy, and radiotherapy.

Adoptive immunotherapy with cytotoxic T lymphocytes (CTLs) reactive with specific viral antigens has proven to be effective. Here, the investigators aim to evaluate the safety and efficacy of multiple infusions of lung cancer specific cytotoxic T lymphocytes cells in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent obtained prior to any study-specific procedures.
2. Age older than 18 years.
3. Patients with refractory, relapsed, metastatic, advanced lung cancer confirmed by histology and biopsy.
4. Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
5. Expected survival ≥ 12 weeks.
6. Not pregnant, and on appropriate birth control if of childbearing potential.
7. Initial hematopoietic reconstitution with

   * neutrophils (ANC) ≥ 1,000/mm^3;
   * platelet (PLT) ≥ 100,000/mm^3.
8. Proper renal and hepatic functions (ULN denotes "upper limit of normal range") with

   * serum creatinine ≤ 2×ULN;
   * serum bilirubin ≤ 2×ULN;
   * AST/ALT ≤ 2×ULN;
   * ALKP ≤ 5×ULN;
   * serum bilirubin. 2.0 is acceptable in the setting of known Gilbert's syndrome.
9. Human immunodeficiency virus (HIV) and Hepatitis C virus (HCV) test were negative.

Exclusion Criteria:

1. Have occurred in 5 years or are currently suffering from other cancers, except for cured cervical cancer, non-melanoma skin cancer and superficial bladder cancer.
2. Previous exposure to mouse CEA antibody.
3. Current or recent treatment (within the 28-day period prior to Day 0) with another investigational drug or previous participation in this study.
4. Minor surgical procedures within 2 days prior to Day 0 (including central venous access device placement for chemotherapy administration, tumor biopsies, needle aspirations).
5. Pregnant or lactating females.
6. Inadequate bone marrow function with

   * absolute neutrophil count < 1,000/mm^3;
   * platelet count < 100,000/mm^3;
   * Hb < 9 g/dL.
7. Inadequate liver and renal function with

   * serum (total) bilirubin > 1.5 x ULN;
   * AST & ALT > 2.5 x ULN (> 5 x ULN in patients with liver metastases);
   * alkaline phosphatase > 2.5 x ULN;
   * serum creatinine >2.0 mg/dl (> 177 μmol/L);
   * urine dipstick for protein uria should be < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hour urine collection and must demonstrate < 1 g of protein/24 hr.
8. Serious active infection requiring i.v. antibiotics at during screening.
9. Subject infected with HCV (HCV antibody positive), HBV (HBsAg positive), HIV (HIV antibody positive), HTLV (HTLV antibody positive), Treponema pallidum antibody positive or TB culture positive.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety of LC-CTLs in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 3 months
  Physiological parameter (measuring cytokine response)

SECONDARY OUTCOMES:
Functional analyses of LC-CTLs in vitro | 2 weeks
  The specificity of LC-CTLs in vitro will be analysed by intracellular cytokine staining (ICCS) or enzyme-linked immunospot assay (ELISPOT).
Anti-tumor effects | 1 year
  Biochemical markers and image scan will be got before and after treatment. Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No